CLINICAL TRIAL: NCT02400047
Title: Dexamethasone, Can it Replace Ketoprofen in the Strategy of Intraoperative Multimodal Analgesia in Paediatric Surgery ? A Prospective Randomized Double-blinded Study. DEXA OP
Acronym: DEXA OP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35RC14_9853_DEXA OP; 2014-005026-35 (EudraCT Number); 141557A-32 (Other: ANSM)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Paediatric surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone 0.2 mg/kg (Experimental): Single injection of DXM (Mylan Dexamethasone® 20 mg/5 ml or 4 mg/1 ml injection ampoule solution) at 0.2 mg / kg after general anesthesia induction and before surgery incision.
  Interventions: Drug: Dexamethasone 0.2 mg/kg
- Dexamethasone 0.4 mg/kg (Experimental): Single injection of DXM (Mylan Dexamethasone® 20 mg/5 ml or 4 mg/1 ml injection ampoule solution) at 0.4 mg / kg after general anesthesia induction and before surgery incision.
  Interventions: Drug: Dexamethasone 0.4 mg/kg
- Ketoprofen 1 mg/kg (Active Comparator): Single injection of ketoprofen (Medac ketoprofen ® 100 mg/4 ml injection ampoule solution) at 1 mg /kg after general anesthesia induction and before surgery incision.
  Interventions: Drug: Ketoprofen 1 mg/kg

INTERVENTIONS:
Drug: Dexamethasone 0.2 mg/kg — Single injection of DXM (Mylan Dexamethasone® 20 mg/5 ml or 4 mg/1 ml injection ampoule solution) at 0.2 mg / kg after general anesthesia induction and before surgery incision.
  Arms: Dexamethasone 0.2 mg/kg
Drug: Dexamethasone 0.4 mg/kg — Single injection of DXM (Mylan Dexamethasone® 20 mg/5 ml or 4 mg/1 ml injection ampoule solution) at 0.4 mg / kg after general anesthesia induction and before surgery incision.
  Arms: Dexamethasone 0.4 mg/kg
Drug: Ketoprofen 1 mg/kg — Single injection of ketoprofen (Medac ketoprofen ® 100 mg/4 ml injection ampoule solution) at 1 mg /kg after general anesthesia induction and before surgery incision.
  Arms: Ketoprofen 1 mg/kg

SUMMARY:
Postoperative pain and nausea-vomiting (PONV) are the first causes of failure in ambulatory care in pediatric surgery. Actually, the paracetamol/ketoprofen combination in intraoperative care is recommended for effective postoperative analgesia in children. However, intravenous ketoprofen doesn't have the marketing authorization for use in children less than 15 years old and its use is mainly justified by the absence of therapeutic alternatives. Recently, findings from published studies suggest that dexamethasone (DXM), which is actually recommended to prevent PONV for children "at risk", at a dose of 0.1mg/kg, would have analgesic properties above 0.15 mg/kg comparable to non-steroidal anti-inflammatories (NSAI).

Main objective :

To examine the effects of intraoperative DXM (0.2mg/kg and 0.4mg/kg) on the intensity of postoperative pain in the post-anaesthetic care unit (PACU) compared to ketoprofen (1mg/kg).

Secondary objectives :

To examine the effects of intraoperative DXM (0.2mg/kg and 0.4mg/kg) compared to ketoprofen (1mg/kg) on the anesthesia emergence delirium, the intensity of postoperative pain, the consumption of rescue analgesics and the side effects in the first 24 hours after surgery.

DETAILED DESCRIPTION:
Methodology :

Non inferiority, phase III, therapeutic trial. Prospective, randomized double-blinded, monocentric study. Inclusion of 567 patients. Inclusion will be performed by the anesthesiologist, the day of surgery during the preoperative visit.

Each patient will be randomised to receive intraoperative DXM (0.2mg/kg), DXM (0.4mg/kg) (max 20mg) or ketoprofen (1mg/kg) (max 100mg).

The clinical data will be collected prospectively in an electronic database. If the hypothesis of non-inferiority is verified, it is planned to test the superiority of the hypothesis secondarily.

Treatment :

Single injection of DXM (Mylan Dexamethasone® 20 mg/5 ml or 4 mg/1 ml injection ampoule solution) at 0.2 mg / kg or 0.4 mg/kg or single injection of ketoprofen (Medac ketoprofen ® 100 mg/4 ml injection ampoule solution) at 1 mg /kg after general anesthesia induction and before surgery incision.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 1 to 16 years
* Undergoing surgery (orchiopexy, inguinal hernia, circumcision, adenoidectomy, tonsillectomy or orthopedic act with osteosynthesis)
* Parental consent

Exclusion Criteria:

* Contraindication to NSAI or DXM
* Hypersensitivity to ketoprofen, DXM, hypnovel or atarax
* Porphyria
* Long QT Syndrome
* Renal or hepatic impairment
* Corticosteroid consumption the week before surgery
* NSAI consumption within 48 hours before surgery
* IV induction for full stomach or myopathic patient.
* French language not spoken by parents.
* Simultaneous participation in biomedical research on health products

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 580 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Maximum intensity of postoperative pain | 1 hour
  Maximum intensity of postoperative pain assessed in PACU using the Faces Legs Activity Cry Consolability tool (FLACC, 0-10)

SECONDARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium Scale (PAEDS) | 24 hours
  Pediatric Anesthesia Emergence Delirium Scale (PAEDS)
Intensity of postoperative pain | 24 hours
  Intensity of postoperative pain assessed in ambulatory unit and at home one day after surgery. (FLACC, 0-10).
Rescue analgesic consumption | 24 hours
  Rescue analgesic consumption in the PACU, ambulatory unit and at home.
Side effects | 24 hours
  Side effects during hospitalization (PONV, postoperative bleeding) and in the first 24 hours post-surgery (PONV, fever, bleeding, behavior modification and sleep disorders).
Length of stay | 24 hours
  Length of stay in ambulatory unit (time of possible discharge using Pediatric Post Anesthetic Discharge Scoring System and the actual time of discharge).
Parent's satisfaction | 24 hours
  Parent's satisfaction on a four-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France